CLINICAL TRIAL: NCT02932878
Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment With DSXS Topical Product in Patients With Plaque Psoriasis
Brief Title: An Open Label, Safety Study to Assess the Potential for Adrenal Suppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSXS 1503a
Record Dates: First submitted 2016-10-12; First posted 2016-10-13 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-11

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSXS topical (Experimental): administered twice daily for 28 days
  Interventions: Drug: DSXS topical

INTERVENTIONS:
Drug: DSXS topical — topical treatment
  Other Names: active

SUMMARY:
An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with DSXS (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

DETAILED DESCRIPTION:
To evaluate the potential of DSXS to suppress HPA axis function in patients with mild to moderate plaque psoriasis.

To evaluate the efficacy parameters and adverse event (AE) profile of DSXS administered to patients with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non pregnant, non lactating females

Exclusion Criteria:

* Patients under 2 years of age

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-02 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novum Pharmaceutical Research Services, Study Chair — http://www.novumprs.com/contact
Locations (1):
- Taro Pharmaceuticals USA Inc., Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DSXS Topical Cohort 1: administered twice daily for 28 days in patients age 12-18 years of age
  DSXS topical: topical treatment
- DSXS Topical Cohort 2: administered twice daily for 28 days in patients age 6-11 years or age
  DSXS topical: topical treatment
Period: Overall Study
Arm/Group | DSXS Topical Cohort 1 | DSXS Topical Cohort 2
Started | 15 | 1
Completed | 13 | 0
Not Completed | 2 | 1
Not completed — Due to Lab Results | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DSXS Topical Cohort 1 | DSXS Topical Cohort 2 | Total
Number analyzed (Participants) | 15 | 1 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.13 (1.88) | 8.00 | 14.69 (2.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 11 | 0 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 12
  Not Hispanic or Latino | 4 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 13 | 1 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Total BSA [Mean (Standard Deviation); unit: meters squared] | 1.86 (0.35) | 1.31 | 1.83 (0.37)
Baseline IGA [Count of Participants; unit: Participants]
  Clear | 0 | 0 | 0
  Minimal | 0 | 0 | 0
  Mild | 7 | 1 | 8
  Moderate | 8 | 0 | 8
  Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients in the Study With HPA Axis Suppression
Description: Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin
Time Frame: 28 Days
Population: The one patient in Cohort 2 did not qualify for evaluation of HPA axis suppression.
Measure: Count of Participants; unit: Participants
Arm/Group | DSXS Topical Cohort 1 | DSXS Topical Cohort 2
Number analyzed (Participants) | 11 | 0
Participants
  Yes | 1 | 0
  No | 10 | 0

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | DSXS Topical Cohort 1 | DSXS Topical Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/1
Other Adverse Events (participants affected / at risk) | 0/15 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/78/NCT02932878/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02932878/SAP_001.pdf